CLINICAL TRIAL: NCT05651282
Title: Uterine Cancer Risk Reducing Strategies in Postmenopausal Women
Brief Title: Risk Evaluation and Screening to Tailor Prevention and Reduce the Incidence of Endometrial Cancer
Acronym: RESToRE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Aline Talhouk, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H22-02290
Record Dates: First submitted 2022-10-11; First posted 2022-12-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Endometrium Cancer
Keywords: Screening; Prevention; Progesterone Challenge Test; Women's Health; Reproductive health; Menopause
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: All eligible participants will move into the various steps of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Progesterone Challenge Test (Experimental): 10-day course of medroxyprogesterone acetate (Provera) 10 mg per os (po) daily.
  Interventions: Drug: Provera

INTERVENTIONS:
Drug: Provera — Progesterone Challenge Test

SUMMARY:
This study proposes to assess feasibility and acceptability of screening and risk reducing interventions in individuals at increased for endometrial cancer (EC). The investigators will use an epidemiological risk model to participants' absolute risk of developing EC in the next 10 years. Those whose absolute risk is 2% or greater or who have a Body Mass Index (BMI) higher than 34.9 will proceed to a second screening test (the Progesterone Challenge Test or the PCT) used to identify those with endometrial proliferation. The PCT consists of taking a ten-day course of medroxyprogesterone acetate (Provera) 10 mg per os daily. If withdrawal bleeding is experienced during the ten days up to two weeks since the final dose, this is considered a positive test result. PCT positive participants will receive standard of care treatment which may include endometrial biopsy and hormone therapy. As part of this project, the investigators will test the utility of self-collected vaginal sampling to measure DNA mutations and microbiome characteristics to help refine who could forego an endometrial biopsy in the future. Participants identified through the PCT will receive a lifestyle intervention through the Small Steps for Big Changes program.

DETAILED DESCRIPTION:
Study Part A

Eligibility Screen 1 - REDCap questionnaire to determine absolute risk of EC: Interested participants will be directed to REDcap where they will provide informed consent for Eligibility Screen 1 and complete a questionnaire with information needed to compute their absolute risk of being diagnosed with EC in the next 10 years. This absolute risk was calculated using the Pfeiffer et al. model (PMID 23935463), and the investigators have defined the threshold of what the investigators consider higher than average risk to be 2%. The investigators have selected this number because the population lifetime risk of EC is 2%; this number also corresponds to a 15% threshold from a similar BC population. For this study any participant whose risk falls above that threshold will be eligible to participate in part B. While this risk score model is not yet validated in the British Columbia population, it considers many factors demonstrated to be highly associated with EC.

Study Part B

1. Invitation to Participate: Participants whose absolute risk is above or equal to 2% will be called by a research coordinator and invited to participate. The investigators anticipate that ~250 high-risk participants will need to be identified for Eligibility Screen 2.
2. Introduction to Primary Care Provider or Gynecologist: A member of the clinical study team will contact the participant's primary care provider to describe the study, inform them of the consent of their patient, and ask the provider if they are willing to participate by prescribing the MPA to the participant and performing any follow up as per standard of care. The primary care provider will also receive a follow-up letter confirming the participant's involvement and summarizing the phone conversation. If the participant has no physician, or if their current primary care provider is unwilling to support them in this study, our clinical study team will help direct them to a local gynaecologist to undergo the PCT and any subsequent standard of care treatment. The only exception to this would be if it was determined that the PCT was medically contraindicated. In this case, the participant would not be able to continue in the study.
3. Appointment for PCT Prescription: Participants will have either a televisit or in-person appointment with their primary care provider or gynaecologist who has agreed to prescribe the 10-day course of MPA (10mg) for the participant to undergo the PCT.
4. At-home Vaginal Swabs and Tampon Collection: Participants who have obtained a prescription for the PCT will be mailed an at-home self-sampling kit for the collection of tampons (only one is required for collection, a spare will be sent in case of error in application) and swabs along with a pH strip and a set of instructions. Participants will be asked to not have sexual intercourse, use vaginal medications, feminine sprays, douches, genital wipes or contraceptive spermicides for 48 hours before providing the self-collection. Participants will be provided with a postage paid return mailing envelope to return the samples to us. Participants will be prompted through MyCap to indicate when they receive their kits, when they complete the self-collection, and when they have mailed back their kits.

   Tampons and swabs will be sent to a Research Coordinator at BC Cancer. Tampons will be processed to extract genetic material, then cell and liquid fractions will also be stored. DNA extractions and targeted sequencing of EC-associated genes will be performed. Tampon and vaginal DNA swabs will be processed and analyzed following the ADVISE study protocols. DNAgenotek OMNIgene vaginal swabs are stable at room temperature for 30 days so will be immediately treated with proteinase K and aliquoted into cryovials for storage at -80C. Samples will be sent to Microbiome Insights for DNA extraction and next- generation sequencing.
5. Eligibility Screen 2 - Progesterone Challenge Test to detect proliferative endometrium: Through the MyCap app, participants will record when they start the PCT. They will receive daily reminders to take the MPA pills and will use the app to identify withdrawal bleeding or any other symptoms. Any participant who is not responsive for two days through the MyCap app will be called by the research coordinator. Those who do not have a smartphone or choose not to use the MyCap, will be managed through email and phone correspondence.

Participants who test positive on the PCT (estimated n~25-50) will receive a phone call from the study coordinator at which time they will be prompted to inform their primary care provider of their withdrawal bleeding and to make a follow-up appointment. They will also be asked to complete a second round of at-home self-collection with vaginal swabs, tampon, and a pH strip.

Simultaneously, a member of our clinical study team will contact the participant's primary care provider to inform them of this positive PCT result, and request that they ensure an appointment is made with this participant. At this time, the clinical study team will also determine who will be performing an endometrial biopsy and where this will occur, as endometrial sampling is standard of care for those who tested positive on PCT. A letter will be sent after this correspondence to all treating physicians for inclusion as part of the patient's records.

7) Return of endometrial biopsy results: The study team will access the biopsy results and any hormonal intervention that may have been prescribed. They will also locate archival material of the endometrial biopsy and request any remaining specimen to be used for translational analysis to be compared to the results from tampon and vaginal swab DNA sequencing.

Study Part C

All participants who complete the PCT will be invited to participate in the final portion of the study.

Lifestyle intervention - The Small Steps for Big Changes (SSBC) program: This is a community-based program for personalized counselling on diet and exercise run by Dr. Mary Jung and her research team at UBC. The program will include six sessions of 1-on-1 exercise and dietary counselling with a trained coach over four weeks (virtually using the University of British Columbia Zoom).

Enrolling in SSBC: The study coordinator will obtain informed consent from any participants who test positive on the PCT and who remain in the study and guide them through next steps involved in the SSBC lifestyle intervention. The study coordinator will mail out a Fitbit, scale and a tape measure to all participants and confirm that the items have been received through MyCap.

Initial Coaching Appointment: A team member from the SSBC program will contact consented participants to schedule their first meeting with a coach. During the first session with the coach, participants will be instructed on how to measure their height, weight, and waist circumference using a tape measure and scale (provided as needed) and they will enter this information on REDCap. In addition, participants will be asked to create their individual health report by completing a survey through REDCap that will ask about physical activity, dietary behaviours, and utilization of healthcare.

Conforming to the SSBC program, the first and second week of the program will include two virtual sessions per week with a coach and three independent exercise sessions that participants are expected to complete on their own each week. The third and fourth week will include one virtual session with a coach and four independent exercise sessions to be completed weekly. Each week the exercise durations will become progressively longer.

Adherence to diet in SSBC is assessed weekly on REDCap using a validated food frequency questionnaire and exercise is assessed via self-report on REDCap.

Follow-up

Lifestyle Intervention: After the initial four weeks of the program, participants will have a check-in with a coach at the 3-month mark to assess progress and adherence to the program.

Exit survey: Participants, depending on the stage at which they exit the study, will be asked about their experience using the MyCap app, and with the at home vaginal sampling kits, the PCT, biopsy, SSBC program, and whether they found these acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Individuals are postmenopausal (must be three (3) years past last menstrual period)
* Individuals have an intact uterus (have not had a hysterectomy)

Exclusion Criteria:

* Individuals taking hormone therapy for menopause (including vaginal estrogen)
* Individuals taking male hormones,
* Individuals on anti-endocrine therapy (such as tamoxifen)
* Individuals on aromatase inhibitor therapy
* Individuals who have experienced abnormal uterine bleeding
* Individuals who have an Intrauterine Device (IUD)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Proposed Screening Method | Through study completion, an average of 1 year
  Feasibility will be measured through rates of study enrollment, drop out, and adherence to intervention protocol. To be considered feasible, the study must meet all three of the following criteria: (1) enrollment and accruals: at least 80% of individuals in the top 30 percentile for risk will agree to and complete the PCT; (2) retention: at least a 50% overall retention rate after eligibility from first screen to 3 months post intervention; (3) adherence: at least 75% of participants compliant with interventions as directed (i.e. participating in at least five of the six SSBC sessions). If either accrual, retention, or adherence criteria is violated, the study will be deemed not feasible.
Acceptability of Proposed Screening Method | Through study completion, an average of 1 year
  Acceptability will be measured through a standardized and validated survey of satisfaction with therapeutic services, the Client Satisfaction Questionnaire-8 (CSQ-8). Acceptability will be defined as a group median score ≥28 (scores range from 8 to 32) on the CSQ-8. Program evaluation items will be analyzed descriptively. The investigators will use analysis of variance to determine whether the feasibility or acceptability varied by social gender, socio demographic, ethnic, age, body size, or geographic location.

SECONDARY OUTCOMES:
Proposed Screening Method Program Evaluation | Through study completion, an average of 1 year
  A secondary measure will be an overall program evaluation which assesses (1) the overall ease of participation and helpfulness of the program, and (2) agreement to a statement about liking the app-based format. This information will be collected through questions asked in an exit survey.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Talhouk, PhD, Principal Investigator — University of British Columbia, Department of Obstetrics and Gynecology; Jessica McAlpine, MD, Principal Investigator — University of British Columbia, Department of Obstetrics and Gynecology
Locations (1):
- VGH Research Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
As per our consent forms IPD is only accessible to PI and research team. De-identified data may be accessible through collaborations.

REFERENCES:
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Obeid JS, McGraw CA, Minor BL, Conde JG, Pawluk R, Lin M, Wang J, Banks SR, Hemphill SA, Taylor R, Harris PA. Procurement of shared data instruments for Research Electronic Data Capture (REDCap). J Biomed Inform. 2013 Apr;46(2):259-65. doi: 10.1016/j.jbi.2012.10.006. Epub 2012 Nov 10. PMID 23149159
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Pfeiffer RM, Park Y, Kreimer AR, Lacey JV Jr, Pee D, Greenlee RT, Buys SS, Hollenbeck A, Rosner B, Gail MH, Hartge P. Risk prediction for breast, endometrial, and ovarian cancer in white women aged 50 y or older: derivation and validation from population-based cohort studies. PLoS Med. 2013;10(7):e1001492. doi: 10.1371/journal.pmed.1001492. Epub 2013 Jul 30. PMID 23935463
- [Background] Hart GR, Yan V, Huang GS, Liang Y, Nartowt BJ, Muhammad W, Deng J. Population-Based Screening for Endometrial Cancer: Human vs. Machine Intelligence. Front Artif Intell. 2020 Nov 24;3:539879. doi: 10.3389/frai.2020.539879. eCollection 2020. PMID 33733200
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370